CLINICAL TRIAL: NCT06194890
Title: The Effect of Diverting Attention Technique on Labor Pain and Satisfaction: Randomized-controlled Study
Brief Title: The Effect of Diverting Attention Technique on Labor Pain and Satisfaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Fatma Yildirim, Dr., Hitit University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hitit_Labor
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): When the patients are admitted, their written consent will be obtained and personal information forms and the Visual Comparison Scale (VAS) pain scale will be applied to all participants. VAS pain scale will be applied to both groups during the active phase of labor with 6-8 cm dilatation and 8-10 cm dilatation phases. At the end of the labor, the "Birth Satisfaction Scale Short Form" will be applied to both groups.
- Intervention group (Experimental): When the patients are admitted, their written consent will be obtained and personal information forms and the Visual Comparison Scale (VAS) pain scale will be applied to all participants.
  Women in the experimental group will watch a 15-20 minute video with comedy content during the active phase of the action (4-6 cm dilation), and no intervention will be made to women in the control group.
  VAS pain scale will be applied to both groups during the active phase of labor with 6-8 cm dilatation and 8-10 cm dilatation phases. At the end of the labor, the "Birth Satisfaction Scale Short Form" will be applied to both groups.
  Interventions: Other: Distraction technique with comedy video

INTERVENTIONS:
Other: Distraction technique with comedy video — Women in the intervention group will watch an average of 6 minutes of comedy videos during the active phase, transition phase and latent phase of labor.
  Arms: Intervention group

SUMMARY:
Having a patient with pain watch a video can be used to "direct attention to a different direction", which is a part of nursing care in pain management (İnal and Canbulat, 2015). There are studies using different non-invasive methods to reduce pain during labor (Ebrahimian and Bilandi, 2021; Kazeminia et al., 2020). However, no randomized controlled study has been found in which comedy videos were watched for labor pain management and birth satisfaction. For this reason, it is planned to investigate the effect of comedy video on pain and birth satisfaction in this study.

DETAILED DESCRIPTION:
Pregnancy and birth represent a major crisis and stressful period in a woman's life. The quality of experiences during birth affects the mother's physical and emotional health, her desire to have another child, and her emotional relationship with the child (Vaziri et al., 2012). It is stated that there are relationships between increased maternal birth satisfaction and the quality of care and birth services provided (Jha et al., 2017). Lack of satisfaction can lead to postpartum depression, breastfeeding disorders, changes in the mother's attitude towards having another child in the future, and subsequent changes at birth with associated disorders (Sayed et al., 2018). The applicability of methods that can alleviate pain during the birth stages can turn birth into a positive and satisfying experience (Kordi et al., 2018). Among these methods, non-drug and supportive treatments can improve the mental and emotional aspects of birth by reducing the severity of pain and fear, reduce the frequency of elective caesarean sections, and increase the statistics of natural birth. Despite treatment measures, when a pregnant woman experiences pain and stress, the sympathetic nervous system is constantly stimulated, resulting in an increase in the secretion of catecholamines and therefore an increase in pulse rate and systolic blood pressure (Makvandi et al., 2013). The increase in catecholamines may reduce blood flow from the mother to the fetus, ultimately causing uterine contractions to be less effective and prolonging labor. Therefore, improving maternal and fetal outcomes is recommended to positively impact maternal satisfaction with birth (Zare et al., 2017).

Measures aimed at reducing pain and shortening the length of labor stages may increase maternal satisfaction with the birth experience ( Kordi et al., 2018 ). Maternal and fetal complications limit the use of pharmacological methods to facilitate birth; For this reason, more user-friendly, non-prescription, lower-cost and less complicated methods are preferred (Mirghafourvand et al., 2014). Although there are many techniques available today to make the birth experience enjoyable, it is still important to find more easily applicable methods (Siddiquee et al., 2016). One of the non-medical interventions to reduce sensitivity is the cognitive-behavioral approach; With this approach, the individual's attention is shifted from a painful stimulus to an external stimulus (Indovina et al., 2016). This non-pharmacological approach can be adopted to alleviate stress and lower cortisol concentrations in response to stress. Having a patient with pain watch a video can be used to "direct attention to a different direction", which is a part of nursing care in pain management (İnal and Canbulat, 2015). There are studies using different non-invasive methods to reduce pain during labor (Ebrahimian and Bilandi, 2021; Kazeminia et al., 2020). However, no randomized controlled study has been found in which comedy videos were watched for labor pain management and birth satisfaction. For this reason, it is planned to investigate the effect of comedy video on pain and birth satisfaction in this study.

ELIGIBILITY:
Inclusion Criteria:

* Being in the active phase of labor,
* Being between the ages of 18-45,
* Knowing Turkish,
* Not having a high-risk pregnancy diagnosis,
* Being over 37 weeks gestational age,
* Volunteering to participate in research.

Exclusion Criteria:

* Not knowing Turkish,
* Being diagnosed with a high-risk pregnancy,
* The gestational age is less than 37 weeks,
* Having passed the active phase of labor or being in the latent phase.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — In the labor
Enrollment: 70 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-02-08 (Estimated); Study Completion 2024-04-08 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | in the labor's 4-6, 6-8,8-10 cm cervical opening
  Visual Analog Scale for labor pain

SECONDARY OUTCOMES:
Birth satisfaction scale | In the 4th stage of labor
  Birth satisfaction scale

CONTACTS AND LOCATIONS:
Locations (1):
- Fatma Yıldırım, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No